CLINICAL TRIAL: NCT05802628
Title: A Single-arm, Open-label Study to Explore the Salivary Concentration of Cetylpyridinium Chloride Buccal Tablets After Single-dose Administration in Healthy Subjects
Brief Title: Salivary Drug Concentration Exploratory Study of Cetylpyridinium Chloride Buccal Tablets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Fang, Professor of Pharmacy, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MLD-C-23001
Record Dates: First submitted 2023-03-26; First posted 2023-04-06 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Pharyngitis Acute; Gingivitis
Keywords: salivary drug concentration
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational group (Experimental)
  Interventions: Drug: Cetylpyridinium Chloride Buccal Tablets

INTERVENTIONS:
Drug: Cetylpyridinium Chloride Buccal Tablets — Subjects administrated single dose of Cetylpyridinium Chloride Buccal Tablet

SUMMARY:
The study is a single-arm, open-label study to explore the salivary concentration of Cetylpyridinium Chloride Buccal Tablets after single-dose administration in Healthy Subjects

DETAILED DESCRIPTION:
Primary Objective: To observe the concentration of the investigational product in the saliva of healthy subjects.

Secondary purpose: To observe the safety of the investigational product in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have fully understand the objective, character, methods and potential adverse reactions of the trial, voluntarily participate in the study, and sign the informed consent form before enrolled into the study.
2. Healthy subjects aged 18-45 (both inclusive) with an appropriate ratio of male to female.
3. Subjects who had no parenthood plan from the signing of the informed consent form to one month after completing study, and agreed to take effective and appropriate contraceptive measures voluntarily by themselves and their partners during this period.
4. Subjects those who be able to communicate well with investigators, and be able to understand and comply with the requirements of this study.

Exclusion Criteria:

1. Allergic to any ingredients of this product or excipients (sucrose, Hypromellose, Carbomer 934P, Tartrazine aluminium lake, menthol,Magnesium octadecanoate, Povidone K 30)
2. Pregnant or breastfeeding women
3. Participants with abnormal salivary secretion, such as patients with xerostomia and diabetic dry mouth
4. Usage of oral stimulants, salivary gland stimulants, other treatments or saliva substitute treatment that may affect salivary gland secretion within 7 days before screening
5. Those who cannot tolerate venipuncture or have a history of haemorrhage or needle fainting
6. Those who on special diet, who cannot comply with the standard diet of the study center, who have difficulty swallowing, who are lactose intolerant, or who have galactosemia or glucose/galactose absorption disorders
7. Those who indicated as abnormal with clinical significance in screening laboratory examination, physical examination, vital signs or electrocardiogram inspection based on judgement of clinical study doctor.
8. The subjects may not be able to complete the study following protocol due to other reasons or investigators judge that they are not suitable participants.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Salivary plasma drug concentration | 15 minutes, 0.5 hour, 1 hour, 1.5 hours, 2 hours after dosing
  Detecting the salivary drug concentration after dosing

SECONDARY OUTCOMES:
Total salivary volume | The total salivary volume at the same time point on Day 0 and Day 1
  Collecting the total salivary volume

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Xie Z, Chen L, Liu X, Li S, Ye S, Tang H, Lee C, Gu Q, Men F, Zhang J, Hu D, Jiang Y, Wang X, Wang Q, Feng Y, Niu S, Liu Y, Fang Y. An exploratory study of drug concentration and inhibitory effect of cetylpyridinium chloride buccal tablets on SARS-CoV-2 infection among 10 Chinese subjects. Fundam Clin Pharmacol. 2024 Jun;38(3):579-587. doi: 10.1111/fcp.12972. Epub 2023 Nov 20. PMID 37985697